CLINICAL TRIAL: NCT05296252
Title: Attention and Achievement (A Subproject Affiliated With the Texas Center for Learning Disabilities or TCLD)
Brief Title: Attention and Achievement: A Mind Wandering Investigation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Houston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 00000568
Record Dates: First submitted 2022-01-25; First posted 2022-03-25 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2022-05

CONDITIONS: Attention Disturbances

STUDY DESIGN:
Intervention Model Description: The factors are study condition order (reading, math), proactive and reactive mind-wandering manipulation (yes, no), and lesson target (reading, math, both, neither)
Masking Description: There is no need, and it is not possible to blind condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mind Wandering Intervention (Experimental): 75% of participants will receive proactive and reactive mind-wandering information and redirection.
  Interventions: Behavioral: mind-wandering intervention
- Mind Wandering Comparison (Active Comparator): 25% of participants will receive only mind-wandering redirection, but only at random times.
  Interventions: Behavioral: mind-wandering comparison

INTERVENTIONS:
Behavioral: mind-wandering intervention — Participants in this condition receive a brief introduction to the potential impact of mind-wandering (before learning, proactive), and are redirected to lesson if "probe-caught" mind-wandering are endorsed (during learning, reactive)
  Arms: Mind Wandering Intervention
Behavioral: mind-wandering comparison — Participants in this condition receive no introduction, and only redirection, and the redirection is random, not in reaction to mind-wandering
  Arms: Mind Wandering Comparison

SUMMARY:
This study assesses the impact of mind-wandering on reading and math.

DETAILED DESCRIPTION:
This study assesses the impact of mind-wandering on reading and math. Specifically 120 middle school student participants will receive descriptive measures (of achievement, attention and related factors including mind-wandering), and will receive a brief (~30 min) lesson in reading and math (order counterbalanced). Participants will receive a brief pre-test, the lesson, and then a post-test on the reading and math outcomes. 75% of the participants will receive a brief manipulation that sets up the influence of mind-wandering, as well as redirects when probe-caught mind-wandering occurs. The remaining participants will receive only redirects, and only randomly. Among participants to receive the mind-wandering manipulation, an equal number will receive this only for reading, only for math, and for both reading and math.

ELIGIBILITY:
Inclusion Criteria:

* enrollment in schools where we have permission to conduct the study

Exclusion Criteria:

* students known to be enrolled in separate curricula (e.g., life-skills classes)

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 53 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Investigator Developed Items Derived From Reading Content Being Taught | administered one time immediately following the single reading learning session on day 1
  Participants will answer multiple choice questions regarding the reading material being taught, and the key index will the raw score number correct. The investigators call the scale "Sleep and Dreams" (after the content the participant is reading about), and the possible score range will be 0 (min) to 24 (max), with higher scores meaning better comprehension of the material.
Investigator Developed Items Derived From Math Content Being Taught | adminstered one time immediately following the single math learning session on day 1
  Participants will answer multiple choice questions regarding the math material being taught, and the key index will the raw score number correct. The investigators call the scale "Circles" (after the content being taught), and the possible score range will be 0 (min) to 24 (max), with higher scores meaning better comprehension of the material.

SECONDARY OUTCOMES:
Investigator Developed Probe-Caught Mind-Wandering | On 12 occasions interspersed during each of the math and reading learning sessions, on day 1 only.
  During the learning (of the reading and math content), participants are prompted on several occasions as to whether their mind was wandering during the lesson. This is a single item multiple/choice scale (called Probe-Caught Mind Wandering), with the range being 0 (min) to 12 (max), with lower scores indicating the better outcome (less mind wandering)

CONTACTS AND LOCATIONS:
Overall Officials: Paul T. Cirino, PhD, Principal Investigator — University of Houston
Locations (1):
- University of Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
If another researcher with an approved Institutional Review Board (IRB) protocol wishes to utilize the data for purposes that are non-overlapping with the investigators, they may reach out to the Study PI, who can share de-identified individual data.
Supporting Information: Study Protocol, ICF
Time Frame: Data will become available after the paper describing the study is published in a peer-reviewed Journal, and will be available for up to 5 years following the termination of the study
Access Criteria: If another researcher with an approved Institutional Review Board (IRB) protocol wishes to utilize the data for purposes that are non-overlapping with the investigators, they may reach out to the Study PI, who can share de-identified individual data.